CLINICAL TRIAL: NCT02486536
Title: The Best Dosage and Timing of PEG for Bowel Preparation Before Capsule Endoscopy a Prospective, Single-Blind, Randomized, Multi-center Study
Brief Title: The Best Dosage and Timing of Polyethylene Glycol for Bowel Preparation Before Capsule Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhizheng Ge (Other)
Collaborators: Huashan Hospital (Other); Shanghai East Hospital (Other); Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhizheng Ge, MD, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2015-045k
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Small Bowel Disease
Keywords: capsule endoscopy; polyethylene glycol; bowel preparation solutions
MeSH Terms: interventions — Polyethylene Glycols; Capsule Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Active Comparator): Fast for 12h before the examination and take 8ml of Simethicone Emulsion (Berlin-Chemie, Germany, containing 40 mg simethicone in 1mL emulsion) with 250ml water 30min before capsule ingestion.CE are performed with the Pillcam SB2 capsule endoscopy system (Given Imaging Co. Ltd., Yoqnem, Israel).
  Interventions: Device: capsule endoscopy
- Group B (Active Comparator): the same as protocol A plus 1L Polyethylene glycol 11-12h before VCE. CE are performed with the Pillcam SB2 capsule endoscopy system.
  Interventions: Drug: polyethylene glycol; Device: capsule endoscopy
- Group C (Active Comparator): the same as protocol A plus 2L Polyethylene glycol 10-12h before VCE. CE are performed with the Pillcam SB2 capsule endoscopy system.
  Interventions: Drug: polyethylene glycol; Device: capsule endoscopy
- Group D (Active Comparator): Group D: the same as protocol A plus 1L Polyethylene glycol 3-4h before VCE. CE are performed with the Pillcam SB2 capsule endoscopy system.
  Interventions: Drug: polyethylene glycol; Device: capsule endoscopy
- Group E (Active Comparator): Group E: the same as protocol A plus 2L Polyethylene glycol 2-4h before VCE. CE are performed with the Pillcam SB2 capsule endoscopy system.
  Interventions: Drug: polyethylene glycol; Device: capsule endoscopy

INTERVENTIONS:
Drug: polyethylene glycol
  Arms: Group B; Group C; Group D; Group E
Device: capsule endoscopy

SUMMARY:
The aim of this study is to evaluate the ideal dose of PEG and timing of bowel preparation in patients referred for CE examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years and referred to capsule endoscopy because of suspected small-bowel disease are prospectively eligible for entry into the study.

Exclusion Criteria:

* Age < 18 or > 75 years
* Known or suspected GI stricture or fistula
* A history of GI tract resection
* Swallowing disorders
* Intensive therapy with fasting and parenteral nutrition;with a disease that may reduce movement of the GI tract, such as diabetes mellitus
* Medications that could affect gastrointestinal movement within one week
* Implanted with a medical electronic device
* Active inflammatory bowel disease, toxic megacolon, toxic colitis
* Severe pulmonary, cardiac, renal, or hepatic disease
* Uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg);
* Disturbance of electrolytes
* Pregnancy or lactation
* Patients inability to provide written voluntary informed consent
* Participation in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
the quality of visualization of the small bowel | one week after CE procedure
  The image quality was evaluated only in cases in which the capsule reached the cecum within the examination period. All CE images will be assessed at low speed (10 frames/s) under the AutoView mode of the RAPID workstation (Given Imaging). The intestinal mucosa is defined as clean if, less than 25% of the mucosal surface was covered by dark liquid, bubbles or debris. Using a timer, the investigators record the exact time period during which the small intestinal mucosa was clean. The definition of "excellent" is at least 90% of the overall small bowel mucosa is clean (the sum of "clean" time /total small bowel transit time>90%). And the definition of "good" is at least 80% of the overall small bowel mucosa is clean. We considered that "excellent" or "good" preparation is adequate to make an accurate diagnosis.

SECONDARY OUTCOMES:
patient acceptability | day of CE procedure
  A visual analogical scale (VAS) is used to evaluate the degree of patients' discomfort. The numerical scale between 0 and 10, with 0 being no burden at all and 10 indicating an intolerable procedure.
  The questionnaire provide information about whether they experienced nausea, bloating, or any discomfort during the bowel preparation, difficulty to complete the preparation, their willingness to repeat the same preparation in the future (yes or no)and did it affect their daily activity and nocturnal rest.
diagnostic rate | one year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Tongren Hospital Affiliated to Shanghai Jiaotong University, China, Shanghai, Shanghai Municipality
  - Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Wu S, Zhong L, Zheng P, Wang YG, Ding WQ, Yu Q, Hui PP, Chen HM, Gao YJ, Ge ZZ. Low-dose and same day use of polyethylene glycol improves image of video capsule endoscopy: A multi-center randomized clinical trial. J Gastroenterol Hepatol. 2020 Apr;35(4):634-640. doi: 10.1111/jgh.14899. Epub 2019 Dec 15. PMID 31682026